CLINICAL TRIAL: NCT00580801
Title: A Phase IIa Randomized, Partially Blinded Trial of Telaprevir (VX-950) in Treatment-Naive Subjects With Chronic Genotype 4 Hepatitis C Infection
Brief Title: An Exploratory Study of Telaprevir in Treatment-Naive Participants With Chronic Genotype 4 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013714; VX-950-TiDP24-C210; NCT00614237 (obsolete NCT alias)
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Telaprevir; Pegylated-interferon-alfa-2a; Pegasys; Ribavirin; Copegus
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telaprevir and then Pegylated-interferon-alfa-2a+Ribavirin (Experimental): Telaprevir 750 milligram (mg) tablet will be administered three times a day orally for 2 weeks and after that pegylated-interferon-alfa-2a (180 microgram [mcg] subcutaneous injection [injected under the skin by way of a needle], once weekly) and ribavirin (1000-1200 mg as oral tablet daily) will be administered from Week 2 to 50.
  Interventions: Drug: Telaprevir; Drug: Pegylated-interferon-alfa-2a; Drug: Ribavirin
- Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin (Experimental): Telaprevir 750 mg tablet will be administered three times a day orally for 2 weeks along with pegylated-interferon-alfa-2a (180 mcg subcutaneous injection, once weekly) and ribavirin (1000-1200 mg as oral tablet daily), from Week 1 to 48.
  Interventions: Drug: Telaprevir; Drug: Pegylated-interferon-alfa-2a; Drug: Ribavirin
- Placebo+Pegylated-interferon-alfa-2a+Ribavirin (Active Comparator): Matching placebo tablet to telaprevir will be administered three times a day orally for 2 weeks along with pegylated-interferon-alfa 2a (180 mcg subcutaneous injection, once weekly) and ribavirin (1000-1200 mg as oral tablet daily), from Week 1 to 48.
  Interventions: Drug: Pegylated-interferon-alfa-2a; Drug: Placebo; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — Telaprevir 750 milligram (mg) tablet will be administered three times a day orally for 2 weeks.
  Arms: Telaprevir and then Pegylated-interferon-alfa-2a+Ribavirin; Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Drug: Pegylated-interferon-alfa-2a — Pegylated-interferon-alfa-2a (180 microgram [mcg] subcutaneous injection, once weekly) will be administered from Week 1 to Week 48 or 50.
Drug: Placebo — Matching placebo tablet to telaprevir was administered three times a day orally for 2 weeks.
  Arms: Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Drug: Ribavirin — Ribavirin (1000-1200 mg as oral tablet daily) will be administered from Week 1 to Week 48 or 50.

SUMMARY:
The purpose of this study is to evaluate the activity and safety of telaprevir on Hepatitis C Virus (HCV) Genotype 4, alone or in combination with standard therapy, that is, pegylated-interferon-alfa-2a and ribavirin in treatment-naive (never been treated before with antiretroviral therapy) participants.

DETAILED DESCRIPTION:
This is a Phase 2a, partially-blind, randomized (study drug assigned by chance) and multiple-dose study to evaluate the activity and safety of telaprevir on HCV early viral kinetics in treatment-naive participants who are chronically infected with HCV Genotype 4. The study consists of 4 parts: Screening period (6-week); Investigational Treatment period (consisting of 2-week treatment with telaprevir or telaprevir+standard treatment or placebo); Standard Treatment period (consists of 46 or 48-week standard treatment); and Follow-up period (24-week). The activity of telaprevir will be evaluated by early viral kinetic parameters along with viral response and pharmacokinetic assessments during the investigational treatment phase. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: - Participant has chronic Genotype 4 Hepatitis C infection

* Plasma hepatitis C virus (HCV) ribonucleic acid (RNA) level greater than 10,000 International unit per milliliter (IU/mL) at Screening
* Participant never received treatment for HCV
* Participant was to be in good health (besides HCV infection), in the opinion of the Investigator, judged on the basis of medical history and physical examination (including vital signs and screening electrocardiogram [ECG]), with any chronic medical conditions under stable medical control
* Participant had to be willing to refrain from the concomitant use of any medications or substances Exclusion Criteria: - Participants with history or evidence of cirrhosis or history of suspicion of alcohol, barbiturate, or amphetamine recreational or narcotic drug use, which in the Investigator's opinion would compromise the participant's safety and/or compliance with study procedures
* Participant has human immunodeficiency virus (HIV) or hepatitis B virus (HBV) co-infection
* Female participants who are pregnant, or planning to become pregnant, or breastfeeding, and partners of female participants who are pregnant or breastfeeding
* Participant has hypersensitivity to tartrazine
* Participant had participated in any clinical trial for an investigational drug within 90 days before drug administration or participated in more than 2 drug studies in the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA

REFERENCES:
- [Derived] De Meyer S, Ghys A, Dierynck I, Beumont M, Luo D, Picchio G. Virologic characterization of genotype 4 hepatitis C virus variants in patients treated with telaprevir. Virol J. 2014 May 16;11:93. doi: 10.1186/1743-422X-11-93. PMID 24886541

RESULTS

PARTICIPANT FLOW:
Groups:
- Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin: Telaprevir 750 milligram (mg) tablet was administered three times a day orally for 2 weeks and after that pegylated-interferon-alfa-2a (180 microgram [mcg] subcutaneous injection [injected under the skin by way of a needle], once weekly) and ribavirin (1000-1200 mg as oral tablet daily) was administered from Week 2 to 50.
- Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin: Telaprevir 750 mg tablet was administered three times a day orally for 2 weeks along with pegylated-interferon-alfa-2a (180 mcg subcutaneous injection, once weekly) and ribavirin (1000-1200 mg as oral tablet daily) was administered from Week 1 to 48.
- Placebo+Pegylated-interferon-alfa-2a+Ribavirin: Matching placebo tablet to telaprevir was administered three times a day orally for 2 weeks along with pegylated-interferon-alfa-2a (180 mcg subcutaneous injection, once weekly) and ribavirin (1000-1200 mg as oral tablet daily) was administered from Week 1 to 48.
Period: Overall Study
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Started | 8 | 8 | 8
Completed | 2 | 7 | 5
Not Completed | 6 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Reached a virologic endpoint | 0 | 1 | 2
Not completed — Participant non-compliant | 0 | 0 | 1
Not completed — Travel | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Median (Inter-Quartile Range); unit: Years] | 43 [36 to 61] | 41 [28 to 52] | 46 [30 to 56] | 45.5 [28 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 5 | 6 | 4 | 15
Region of Enrollment [Number; unit: Participants] — All Participants enrolled were from France.
  Participants
    France | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at Day 15
Description: The plasma HCV RNA levels were used to assess the antiviral activity which included viral response as either undetectable HCV RNA (that is no HCV target was detected in the plasma sample) or less than 25 International unit per milliliter (IU/mL) of HCV RNA (that is Plasma sample contained HCV RNA at a concentration below the limit of quantification [LLOQ=25 IU/mL] of the viral load assay). Plasma HCV RNA levels were measured using the COBAS TaqMan HCV test Version 2.0. This assay used real-time reverse transcription-polymerase chain reaction (RT-PCR) methodology.
Time Frame: Baseline and Day 15
Population: Full analysis included all randomized participants who received at least one dose of the telaprevir or placebo. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Median (Full Range); unit: log 10 IU/mL
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8 | 8
log 10 IU/mL
  HCV RNA levels: Baseline (n=8,8,8) | 5.83 [5.2 to 6.5] | 6.16 [5.4 to 6.8] | 5.88 [5.0 to 6.8]
  HCV RNA levels: Change at Day 15 (n=7,8,8) | -0.77 [-2.9 to 0.3] | -4.32 [-5.2 to 0.0] | -1.58 [-4.0 to -0.8]

2. Secondary Outcome: Percentage of Participants With Viral Response (Undetectable HCV RNA)
Description: Viral response was either defined as having undetectable HCV RNA (that is, no HCV RNA was detected in the participants' plasma samples) or less than 25 IU/mL HCV RNA from Day 15 up to end of treatment (EOT), that is Week 48/50 or early discontinuation. In Week x/y, where, x represents time frame for Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin and Placebo+Pegylated-interferon-alfa-2a+Ribavirin and; y represents time frame for Telaprevir and Pegylated-interferon-alfa-2a+Ribavirin treatment group.
Time Frame: Day 15 up to EOT (Week 48/50 or early discontinuation)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8 | 8
Percentage of participants
  Day 15 (n=7, 8, 8) | 0 | 12.5 | 0
  Week 4/6 (n=7, 8, 8) | 42.9 | 37.5 | 12.5
  Week 12/14 (n=7, 8, 7) | 85.7 | 75.0 | 57.1
  Week 24/26 (n=6, 8, 8) | 100 | 87.5 | 62.5
  Week 36/38 (n=6, 8, 5) | 100 | 75.0 | 100
  Week 48/50 (n=4, 7, 5) | 100 | 85.7 | 100
  EOT (n=8, 8, 8) | 87.5 | 75.0 | 75.0

3. Secondary Outcome: Median Time to First Viral Response (Undetectable HCV RNA)
Description: Time to first viral response (Undetectable HCV RNA) is defined as the number of days since the start of study medication until first time negative HCV RNA level that is less than 25 IU/mL was detected.
Time Frame: Up to Week 48/50
Population: Full analysis included all randomized participants who received at least one dose of the telaprevir or placebo.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8 | 8
Days | 93 [44 to 100] | 85.50 [29 to 171] | 128 [86 to 200]

4. Secondary Outcome: Number of Participants With Viral Breakthrough (Detectable HCV RNA)
Description: Viral breakthrough was defined as having a confirmed increase greater than 1 log 10 in HCV RNA level from the lowest level reached, or a confirmed level of HCV RNA greater than 100 IU/mL in participants whose HCV RNA had previously become undetectable [less than 25 IU/mL]). In Week x/y, where, x represents time frame for Telaprevir+pegylated-interferon-alfa-2a+Ribavirin and Placebo+pegylated-interferon-alfa-2a+Ribavirin and y represents time frame for Telaprevir and then Pegylated-interferon-alfa-2a+Ribavirin treatment group.
Time Frame: Day 8, Day 12, Day 15, Week 24/26 and Week 36/38
Population: Full analysis included all randomized participants who received at least one dose of the telaprevir or placebo.
Measure: Number; unit: Participants
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Day 8 | 1 | 0 | 0
  Day 12 | 3 | 0 | 0
  Day 15 | 5 | 0 | 0
  Week 24/26 | 5 | 0 | 1
  Week 36/38 | 5 | 2 | 1

5. Secondary Outcome: Percentage of Participants With Sustained Viral Response (SVR)
Description: Sustained viral response was defined as having undetectable HCV RNA at EOT (Week 48/50 or early discontinuation) and no confirmed detectable HCV RNA levels between EOT and 12 weeks (SVR12) and 24 weeks (SVR24) after the last dose of study medication.
Time Frame: Week 12 and 24 after the last dose of study medication
Population: Full analysis included all randomized participants who received at least one dose of the telaprevir or placebo.
Measure: Number; unit: Percentage of participants
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8 | 8
Percentage of participants
  SVR12 | 75.0 | 50.0 | 62.5
  SVR24 | 62.5 | 50.0 | 62.5

6. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as having confirmed detectable HCV RNA during the 24-week follow-up period in participants who had undetectable HCV RNA at EOT (Week 48/50 or early discontinuation). Participants who dropped out between 24-week follow-up after EOT were not evaluated for relapse.
Time Frame: Week 24 after EOT (Week 48/50 or early discontinuation)
Population: Full analysis included all randomized participants who received at least one dose of the telaprevir or placebo. "N" signifies those participants who were evaluated for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 7 | 6 | 6
Percentage of participants | 14.3 | 33.3 | 16.7

7. Secondary Outcome: Area Under the Serum Concentration-Time Curve (AUC)
Description: The AUC is a measure of the serum concentration-time curve, calculated by the lin-up/log-down method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose on Day 1 and 15
Population: Intent-to-treat (ITT) population included any randomized participant who received at least 1 dose of telaprevir/placebo. "n" signifies number of participants with data for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8
nanogram*hour/milliliter (ng*h/mL)
  AUC : Day 1 (n=8, 7) | 6702 (3284) | 7467 (4684)
  AUC : Day 15 (n=7, 7) | 17120 (3599) | 23320 (7065)
Statistical Analysis 1: Comparison: Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin vs Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin; Test type: Superiority or Other; Least square mean ratio = 0.98, 90% CI [0.54 to 1.78] — Day 1: The least square (LS) means of the primary parameters for the test and the reference groups were estimated with a linear mixed effects model controlling for treatment group as fixed effects
Statistical Analysis 2: Comparison: Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin vs Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin; Test type: Superiority or Other; Least square mean ratio = 1.33, 90% CI [1.03 to 1.72] — Day 15: The LS means of the primary parameters for the test and the reference groups were estimated with a linear mixed effects model controlling for treatment group as fixed effects

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of Telaprevir
Description: The Cmax is the maximum observed serum concentration, which was measured at Day 1 and 15 for telaprevir and then pegylated-interferon-alfa-2a+Ribavirin (reference) and telaprevir+pegylated-interferon-alfa-2a+Ribavirin (test).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose on Day 1 and 15
Population: ITT population included any randomized participant who received at least 1 dose of telaprevir/placebo. "n" signifies number of participants with data for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8
Nanogram/milliliter (ng/mL)
  Cmax: Day 1 (n=8, 8) | 1598 (803.1) | 1709 (1017)
  Cmax: Day 15 (n=7, 7) | 2733 (554.9) | 3669 (1017)
Statistical Analysis 1: Comparison: Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin vs Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin; Test type: Superiority or Other; Least square mean ratio = 1.00, 90% CI [0.58 to 1.72] — Day 1: The LS means of the primary parameters for the test and the reference groups were estimated with a linear mixed effects model controlling for treatment group as fixed effects
Statistical Analysis 2: Comparison: Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin vs Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin; Test type: Superiority or Other; Least square mean ratio = 1.32, 90% CI [1.05 to 1.66] — [estimate comment as in outcome 7, analysis 2]

9. Secondary Outcome: Pre-Dose Serum Concentration (C[0h]) of Telaprevir
Description: The C(0h) is the pre-dose serum concentration of telaprevir and then pegylated-interferon-alfa-2a+Ribavirin (reference) and telaprevir+pegylated-interferon-alfa-2a+Ribavirin (test).
Time Frame: 0 hour (pre-dose) at Day 15
Population: ITT population included any randomized participant who received at least 1 dose of telaprevir/placebo. "N" signifies those participants who were evaluated for this measure.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 6 | 5
Nanogram/milliliter (ng/mL) | 1873 (376.6) | 2806 (1056.0)
Statistical Analysis 1: Comparison: Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin vs Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin; Test type: Superiority or Other; Least square mean ratio = 1.43, 90% CI [1.02 to 2.02] — [estimate comment as in outcome 7, analysis 2]

10. Secondary Outcome: Minimum Serum Concentration (Cmin) of Telaprevir on Day 15
Description: The Cmin is the minimum serum concentration between 0 hour and τ (τ=dosing interval) of telaprevir and then pegylated-interferon-alfa-2a+Ribavirin (reference) and telaprevir+pegylated-interferon-alfa-2a+Ribavirin (test). Cmin on Day 15 is reported here.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose on Day 15
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 7 | 7
Nanogram/milliliter (ng/mL) | 1639 (447.7) | 2100 (796.3)
Statistical Analysis 1: Comparison: Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin vs Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin; Test type: Superiority or Other; Least square mean ratio = 1.24, 90% CI [0.88 to 1.74] — [estimate comment as in outcome 7, analysis 2]

11. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) of Telaprevir
Description: The tmax is the time to reach maximum observed serum concentration of telaprevir and then pegylated-interferon-alfa-2a+Ribavirin (reference) and pegylated-interferon-alfa-2a+Ribavirin (test).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose on Day 1 and 15
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 8 | 8
Hours
  tmax: Day 1 (n=8, 8) | 4.02 (447.7) [3.00 to 5.97] | 4.00 (796.3) [3.00 to 6.00]
  tmax: Day 15 (n=7, 7) | 2.92 [0.00 to 4.08] | 3.00 [1.92 to 4.00]

12. Secondary Outcome: Average Steady-State Serum Concentration (Css,av) of Telaprevir
Description: The Average steady-state serum concentration (Css,av) was calculated by AUC/τ at steady-state (τ=dosing interval) of telaprevir and then pegylated-interferon-alfa-2a+Ribavirin (reference) and telaprevir+pegylated-interferon-alfa-2a+Ribavirin (test).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose on Day 1 and 15
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin
Number analyzed (Participants) | 7 | 7
Nanogram/milliliter (ng/mL) | 2141 (438.5) | 2896 (842.0)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin | Placebo+Pegylated-interferon-alfa-2a+Ribavirin
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin (N=8) | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin (N=8) | Placebo+Pegylated-interferon-alfa-2a+Ribavirin (N=8)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir and Then Pegylated-interferon-alfa-2a+Ribavirin (N=8) | Telaprevir+Pegylated-interferon-alfa-2a+Ribavirin (N=8) | Placebo+Pegylated-interferon-alfa-2a+Ribavirin (N=8)
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 0
Influenza like illness (General disorders) | 3 | 7 | 4
Asthenia (General disorders) | 0 | 6 | 3
Malaise (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees that before he/she publishes any results of this trial he/she shall allow at least 45 days for the Sponsor to review the pre-publication manuscript prior to submission of the manuscript to the Publisher. In accordance with generally recognized principles of scientific collaboration, co-authorship with any company personnel will be discussed and mutually agreed upon before submission of the manuscript to the Publisher.